CLINICAL TRIAL: NCT01862952
Title: Continuous Video- EEG Monitoring in the Acute Phase in Patients With a Cerebrovascular Attack- Randomisation of a Subpopulation Regarding Treatment Strategy
Acronym: Video-EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC/2013/211
Record Dates: First submitted 2013-05-14; First posted 2013-05-27 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2018-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- antiepileptic treatment as used in daily clinical practice (Active Comparator): Antiepileptic treatment as used in daily clinical practice.
  Interventions: Other: starting of anti-epileptic drug treatment
- No medication (No Intervention)

INTERVENTIONS:
Other: starting of anti-epileptic drug treatment
  Arms: antiepileptic treatment as used in daily clinical practice

SUMMARY:
Stroke is a major cause of epilepsy. The pathophysiological mechanisms of poststroke epilepsy are not known. Subclinical epileptiform discharges could contribute to the neuronal damage and influence functional outcome. Electro-encefalography (EEG) is the golden standard to detect interictal, ictal and subclinical epileptic brain activity.

Patients admitted to the stroke unit with an ischemic or hemorrhagic cerebrovascular attack will undergo a 24 hours video-EEG monitoring to detect epileptiform discharges. Clinical and paraclinical (imaging, serum markers of neuronal damage) parameters will be analysed together with the EEG results. The EEG results will be correlated with the occurence of epileptic seizures and functional outcome and mortality in the acute phase and in the long-term. When subclinical epileptic discharges are found on the EEG, patients will be asked to participate in a second part of the study where they will be randomised into a treatment (with an anti-epileptic drug) versus no-treatment group for a period of 6 months. Outcome parameters will be the occurrence of epileptic seizures, mortality and functional outcome.

Our main hypothesis is that the occurrence of subclinical epileptiform discharges during the acute phase following stroke influences functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic arteria cerebri media infarct and spontaneous intraparenchymal bleeding

Exclusion Criteria:

* Patients with subarachnoidal haemorrhage, traumatic haemorrhage (epidural/subdural bleeding), cerebral venous sinus thrombosis, epilepsy, anti-epileptic treatment, transient ischemic attack, indication for urgent neurosurgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome | day 7
  Modified ranking scale and NIHSS
Functional outcome | at month 6
  Modified ranking scale and NIHSS

SECONDARY OUTCOMES:
Mortality | at month 6
  medical records, seizure diary, interrogation of patient and caregiver
occurrence of epileptic seizures | at month 6
  medical records, seizure diary, interrogation of patient and caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Veerle De Herdt, MD, Phd, Principal Investigator — Ghent University Hospital, Department of Neurology
Locations (1):
- Ghent University Hospital, Ghent, Belgium